CLINICAL TRIAL: NCT01858324
Title: Evaluation of Educational Tools Concerning Hypertension in Ambulatory Pregnant Women, Compared With Usual Antenatal Care
Brief Title: Evaluation of Educational Tools for Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Nadine Sauvé, Member of the Mother & Child Research Axis of the clinical research center Etienne Le Bel, Université de Sherbrooke
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-025
Record Dates: First submitted 2013-05-14; First posted 2013-05-21 (Estimated); Last update posted 2014-12-04 (Estimated); Status verified 2014-12

CONDITIONS: Preeclampsia
Keywords: Preeclampsia; Hypertensive disorders of pregnancy; Patient education; Educationnal tools; Pamphlet; Video; Knowledge; Anxiety; Satisfaction
MeSH Terms: conditions — Pre-Eclampsia; Anxiety Disorders; Personal Satisfaction | interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- educational tools (Experimental): Subjects will receive at time 0 the educational tools (pamphlet-including a graphic-based summary, a magnet and a 12 minutes video). They will then have to answer a questionnaire 1 month later about knowledge, anxiety and satisfaction.
  Interventions: Other: Educational tools
- Usual antenatal care (No Intervention): Subjects in this group will not receive any more educational tools that what is generally offered in routine antenatal care.

INTERVENTIONS:
Other: Educational tools — Subjects will receive the educational tools. They will then receive one month after a questionnaire about knowledge, anxiety and satisfaction.
  Other Names: Pamphlet (including a graphic-based summary); Magnet-summary; Video
  Arms: educational tools

SUMMARY:
Hypertensive disorders of pregnancy happen in 5% of pregnancies. Being aware of symptoms and complications may help women to present early and preserve their own and their baby's health.

The proposed research aims to evaluate the impact of educational tools in pregnant women from an ambulatory population. These tools include a detailed pamphlet (including a graphic-based summary), a magnet summarizing symptoms and appropriate action, and a video. Level of knowledge will be evaluated after one month with a validated questionnaire. We will also evaluate if getting more information about preeclampsia increases patient anxiety as well as satisfaction about the tools.

DETAILED DESCRIPTION:
Background: Preeclampsia is a leading cause of maternal/fetal morbidity/mortality. Pregnant women are often poorly informed on preeclampsia and seeking care too late results in maternal/fetal complications. Many healthcare providers believe that delivering information for low-risk women only make them more anxious.

Preliminary data: We published that an information pamphlet on preeclampsia increases knowledge, without increasing anxiety, and generates high satisfaction in women hospitalized for preeclampsia.

Objectives: Demonstrate that (1) ambulatory low-risk pregnant women will benefit from the pamphlet/video with improved knowledge; (2) without any increase in anxiety, and with great satisfaction.

Design: Prospective randomized controlled pilot study. Inclusion criteria: consecutive pregnant women aged ≥18 y.o. between 200-326 weeks presenting at the clinic and who read/write French or English. Exclusion criteria: Anticipated delivery or termination within one month. Intervention: pamphlet, magnet and video. Control: no educational tool. At baseline, women in both groups will answer questionnaire #1 on demographics; one month later: self-administered questionnaire #2 on knowledge, anxiety, satisfaction.

Sample size: N=178 will provide 80% power to find a significant improvement of at least 20% in knowledge score and 96% power to find a difference of at least 1 on scale for anxiety (alpha of 5%). Assuming a drop-out rate of 10%, missing answers <20%, and rate of answered questionnaire #2 of 50%, 400 subjects will be recruited.

Anticipated results: The tools will improve knowledge by about 20% in intervention group compared to control group. They will not increase anxiety over one point and will be highly appreciated by women.

ELIGIBILITY:
Inclusion Criteria:

* Women between 20+0 to 32+6 weeks pregnant
* Aged 18 years old or more
* Who present at the Blood Sampling in Pregnancy clinic
* With an adequate understanding of written and spoken French or English in order to read the pamphlet and fill out the self-administered questionnaire

Exclusion Criteria:

* Consideration of an interruption of pregnancy for maternal or fetal reasons
* Anticipated delivery within the next month.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2014-03; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Knowledge about preeclampsia | 1 month
  Through a questionnaire (7 questions, 35 statements, one global score)

SECONDARY OUTCOMES:
Anxiety | 1 month
  Question 1: 8 statements (Likert's scale 1 to 6) Question 2 more general
Satisfaction | 1 month
  3 questions

OTHER OUTCOMES:
Sub-group analysis: age | 1 month
  Diferences in outcomes between control and intervention groups according to group age
Sub-group analysis: parity | 1 month
  Differences between control and intervention group according to parity.
Sub-group analysis: pre-pregnancy BMI | 1 month
  Differences between control and intervention group according to pre-pregnancy BMI
Sub-group analysis: category of health care provider | 1 month
  Differences between control and intervention group according to category of healthcare provider
Sub-group analysis: preeclampsia risk factors | 1 month
  Differences between control and intervention group according to preeclampsia risk factors (pre-pregnancy diseases or a history of preeclampsia
Sub-group analysis: tobacco use | 1 month
  Differences between control and intervention group according to tobacco use
Sub-group analysis: | 1 month
  Differences between control and intervention group according to employment type
Sub-group analysis: ethnicity | 1 month
  Differences between control and intervention group according to ethnicity
Sub-group analysis: socio-economic level | 1 month
  Differences between control and intervention group according to socio-economic level
Sub-group analysis: educational level | 1 month
  Differences between control and intervention group according to educational level
Sub-group analysis: marital status | 1 month
  Differences between control and intervention group according to marital status
Sub-group analysis:video viewed on site vs. at home | 1 month
  Differences between control and intervention group according to video viewed on-site vs. at home
Sub-group analysis:delay since last consultation of the tools | 1 month
  Differences between control and intervention group according to delay since last consultation of the tools.

CONTACTS AND LOCATIONS:
Overall Officials: Nadine Sauve, MD, Principal Investigator — Centre de recherche clinique of the Centre Hopitalier Universitaire de Sherbrooke
Locations (1):
- Centre Hopitalier Universiatire de Sherbrooke, Sherbrooke, Quebec, Canada